CLINICAL TRIAL: NCT07049146
Title: Efficacy and Safety of Contrast Endoscopic Ultrasound-Guided Tissue Glue/Coil Devascularization vs. Balloon-Occluded Retrograde Transvenous Obliteration for Preventing Recurrent Gastric Variceal Bleeding: A Prospective Randomized Controlled Trial
Brief Title: Efficacy and Safety of Contrast EUS-Guided Tissue Glue/Coil Devascularization vs. BRTO for Preventing Recurrent Gastric Variceal Bleeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yang Jinlin, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025 Audit No. 670
Record Dates: First submitted 2025-06-10; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Gastric Varices Bleeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided tissue glue/coil injection arm (Experimental): Under linear array endoscopic ultrasound (EUS), puncture GVs with a 19G/22G needle, deploy coils, and inject 1-2ml tissue glue until blood flow in GVs disappears (or inject glue directly if coils are unsuitable). Treat moderate-to-severe esophageal varices (EVs) with band ligation during or after the procedure.
  Interventions: Procedure: EUS-guided tissue glue/coil injection
- BRTO arm (Active Comparator): Establish vascular access via the femoral or internal jugular vein, occlude gastrorenal shunts with a balloon catheter, and inject sclerosant foam. Treat moderate-to-severe EVs with band ligation within 5 days post-procedure.
  Interventions: Procedure: BRTO

INTERVENTIONS:
Procedure: EUS-guided tissue glue/coil injection — Under linear array endoscopic ultrasound (EUS), puncture GVs with a 19G/22G needle, deploy coils, and inject 1-2ml tissue glue until blood flow in GVs disappears (or inject glue directly if coils are unsuitable). Treat moderate-to-severe esophageal varices (EVs) with band ligation during or after the procedure.
  Arms: EUS-guided tissue glue/coil injection arm
Procedure: BRTO — Establish vascular access via the femoral or internal jugular vein, occlude gastrorenal shunts with a balloon catheter, and inject sclerosant foam. Treat moderate-to-severe EVs with band ligation within 5 days post-procedure.
  Arms: BRTO arm

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of EUS-guided tissue glue/coil injection and BRTO in preventing rebleeding of gastric varices (GVs) in patients with portal hypertension and GVs (including those with esophageal varices, ascites, or hepatic encephalopathy). The main questions it aims to answer are:

Is the 1-year all-cause rebleeding rate of EUS-guided tissue glue/coil injection for GVs non-inferior to that of the BRTO group? Does EUS-guided tissue glue/coil injection differ from BRTO in the incidence of decompensated portal hypertension events (variceal bleeding, overt hepatic encephalopathy, ascites) and survival rate post-treatment?

Researchers will compare patients randomized 1:1 to the EUS-guided tissue glue/coil injection arm vs. the BRTO arm to see if there are differences in rebleeding rates and complications.

Participants will:

Receive EUS-guided tissue glue/coil injection or BRTO. Take carvedilol long-term (if no contraindications) to reduce portal pressure. Undergo follow-up assessments at 1, 3, 6, and 12 months ±7 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old;

  * Liver cirrhosis (diagnosed by imaging, laboratory tests, clinical symptoms, or liver biopsy);

    * Experienced bleeding of gastroesophageal varices (GVs) (GOV1, GOV2, or IGV1) within 5 days to 1 year (bleeding lesions observed under endoscopy originating from GVs, or no other bleeding lesions except GVs were found);

      * Presence of spontaneous portosystemic shunts that are technically feasible for BRTO; ⑤ Willing to participate in this clinical study, comply with the study requirements, and sign the informed consent form.

Exclusion Criteria:

* Previously received vascular interventional therapy for preventing rebleeding of GVs;

  * Eligible for variceal ligation treatment of GOV1;

    * Non-cirrhotic portal hypertension (including regional portal hypertension);

      * Previously underwent surgical and interventional shunt procedures;

        * Presence of contraindications to endoscopic or interventional treatment; ⑥ Extensive portal vein thrombosis, cavernous transformation of the portal vein;

          ⑦ Massive ascites;

          ⑧ Concurrent advanced liver cancer or other malignant tumors with a predicted lifespan of less than 3 months;

          ⑨ Concurrent severe diseases of other organs such as the heart, lungs, and kidneys;

          ⑩ Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
One-year all-cause rebleeding rate | one year
  The rate of upper gastrointestinal bleeding occurring within one year after the operation, regardless of the cause

CONTACTS AND LOCATIONS:
Locations (1):
- 37 Guoxue Lane, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No